CLINICAL TRIAL: NCT03216408
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase III Study to Evaluate the Efficacy and Safety of NEURONOX® vs. BOTOX® in Patients With Moderate to Severe Glabellar Lines
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Neuronox and Botox With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG1220MED
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronox (Experimental): Botulinum toxin type A for Injection
  Interventions: Drug: Neuronox
- Botox (Active Comparator): Botulinum toxin type A for Injection
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Neuronox
  Other Names: Clostridium Botulinum Toxin A 100 U
  Arms: Neuronox
Drug: Botox
  Other Names: Clostridium Botulinum Toxin A 50 U
  Arms: Botox

SUMMARY:
This clinical study evaluates the efficacy and safety of Neuronox compared with Botox in adults with moderate to severe glabellar lines.

DETAILED DESCRIPTION:
Subjects are randomly assigned into the two groups at the ratio of 2:1. The purpose of study is to confirm the non-inferiority of Neuronox to Botox in terms of the efficacy and safety in subjects with moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 65
* Subjects with more than grade 2 (moderate) in the investigator's rating of the severity of glabellar lines at maximum frown

Exclusion Criteria:

* Subjects with medical conditions who may be greater risk due to the administration of the investigational drugs
* Subjects with skin disorders at the injection site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
4-grade scale by live assessment of glabellar line severity | 4 weeks after injection
  Glabellar line improvement rate at maximum frown

IPD SHARING:
Plan to Share IPD: Undecided